CLINICAL TRIAL: NCT04795947
Title: Correlation Between Thyroid Function and Quality of Life in Well-controlled Hypothyroidism Patients
Brief Title: Correlation Between Thyroid Function and Quality of Life in Hypothyroidism
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Guang Wang, Director of Endocrinology, Beijing Chao Yang Hospital
Other Study IDs: 2021-PRO39-Hypothyroidism
Record Dates: First submitted 2021-03-10; First posted 2021-03-12 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Hypothyroidism
Keywords: Hypothyroidism
MeSH Terms: conditions — Hypothyroidism

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Behavioral — There is no intervention in this study

SUMMARY:
According to the prevalence survey of thyroid diseases in ten cities in China in 2010, TSH>4.2 mIU /L was the diagnostic cut-off point, and the prevalence of hypothyroidism was 17.8%, including 1.1% clinical hypothyroidism.The annual incidence of hypothyroidism in China is 2.9‰, and primary hypothyroidism is the most common.Typical patients have chilliness, fatigue, swelling of hands and feet, lethargy, memory loss, hypoperspiration, joint pain, weight gain, constipation, menstrual disorder or menorrhagia, infertility, which affects the physiological and psychological functions of patients and reduces the quality of life of patients.The treatment goal of primary clinical hypothyroidism is that the symptoms and signs of hypothyroidism disappear, and TSH, TT4 and FT4 values remain in the normal range.Levothyroxine (L-T4) is the main alternative therapy for this disease.Thyroid disease patients quality of life questionnaire (Thyroid - specific Patient Reported Outcome, ThyPRO) for the development of the Danish scholars such as WATT first can be applied to various comprehensive scale of benign Thyroid disease patients, applied in the Danish people has good reliability and validity, has been translated into ten languages application in many countries the crowd, WATT et al in 2015 developed the scale of the concise version (ThyPRO39).Studies have shown that in the treatment of patients with thyroid disease, even if thyroid function is within the normal range, there are still physiological or psychological impairments such as chills, fatigue, anxiety, depression, which reduces the quality of life of patients.Studies have shown that TSH level in patients with hypothyroidism is correlated with patients' quality of life. Even within the normal range, the higher TSH level is, the worse the patients' quality of life score is, and there is an independent correlation in fatigue and emotional susceptibility.

This study except for other factors, such as merger disease with primary hypothyroidism patients quality of life assessment, observe the normal JiaJian patients, we use the current widely used thyroid disease patients to evaluate the quality of life questionnaire (ThyPRO - 39), observe thyroid hormone levels in patients with hypothyroidism and their quality of life scale and the relevance of the blood sugar, blood lipid metabolic indicators related to relevance.

DETAILED DESCRIPTION:
Hypothyroidism is a systemic metabolic syndrome caused by reduced thyroid hormone production and secretion or reduced tissue function.According to the prevalence survey of thyroid diseases in ten cities in China in 2010, TSH>4.2 mIU /L was the diagnostic cut-off point, and the prevalence of hypothyroidism was 17.8%, of which the prevalence of subclinical hypothyroidism was 16.7%, and the prevalence of clinical hypothyroidism was 1.1% [6].The prevalence was higher in females than in males and increased with age.The annual incidence of hypothyroidism in China is 2.9‰[7].Epidemiological evidence suggests that hypothyroidism is associated with anxiety and mood disorders [4].Several studies have shown that hypothyroidism is associated with lower quality of life (QOL), higher load symptom, poorer physical and mental health, and poorer attention performance.The treatment goal of primary clinical hypothyroidism is that the symptoms and signs of hypothyroidism disappear, and TSH, TT4 and FT4 values remain in the normal range.Levothyroxine (L-T4) is the main alternative therapy for this disease [8].Thypro questionnaire (Thypro) is the first comprehensive scale developed by Danish scholar Watt et al., which is applicable to patients with various benign Thyroid diseases. It has been translated into 10 languages and applied in populations in many countries.[9].Studies have shown that, in the treatment of hypothyroidism patients, even if thyroid function is in the normal range, there are still chills, fatigue, anxiety, depression and other physiological or psychological damage, reducing the quality of life of patients.The relationship between thyroid hormone levels and quality of life in patients with treated hypothyroidism is controversial.Studies have shown that in patients with primary hypothyroidism, higher TSH values are associated with impaired quality of life, even if TSH is within the normal reference range.TSH was positively correlated with the scores of fatigue and emotional susceptibility scales, indicating that these two aspects of quality of life were significantly affected with the increase of TSH level [1].However, some studies have shown that the quality of life of hypothyroidism patients treated with levothyroxine has nothing to do with the level of thyroid hormone, and TSH or free T4 cannot be used as the indicator of the best treatment effect, because it cannot reflect the patient's quality of life [2].But in the study, a significant percentage of patients with hypothyroidism simultaneously with high blood pressure, diabetes, dyslipidemia, diseases such as depression or anxiety, long-term use may affect the metabolism of thyroid hormones and drugs, and combined with the disease itself also has effect on the quality of life in patients with [2], not real thyroid hormone levels in patients with quality of life, their metabolism and the influence of correlation, etc.

This study except for other factors, such as merger disease with primary hypothyroidism patients quality of life assessment, observe the normal JiaJian patients, we use the current widely used thyroid disease patients to evaluate the quality of life questionnaire (ThyPRO - 39), observe JiaJian thyroid hormone levels in patients with son and their quality of life scale and the relevance of the blood sugar, blood lipid metabolic indicators related to relevance.

Signed in patients voluntary and informed consent, to assess all criteria of patients, collected demographic data (such as gender, age, etc.), record the history and the other previous medical history, family history, related to the vital signs data (such as height, weight, waist circumference, hip circumference, BMI and waist hip ratio, blood pressure), laboratory indexes (including thyroid function, HbA1c, fasting insulin, fasting C peptide, blood biochemistry), thyroid ultrasound.Patients meeting the inclusion criteria received two questionnaires: ThyPRO-39 (Chinese version), and the MOS 36-item Short Form Health Survey (SF36).ThyPRO39 has 39 items, 12 subscale tables and 1 single item to evaluate overall quality of life.The 12 subscales were further divided into 3 categories: (1) somatic symptoms (goiter symptoms, hyperthyroidism symptoms, hypothyroidism symptoms, thyroid ophthalmopathy symptoms);(2) physiological (fatigue, cognition), psychological (anxiety, depression, mood) and social (social activities, daily life);(3) the appearance.This scale is a self-rating scale, and Likert 5-grade score is used to calculate the crude score of each subscale, and then the control scoresheet and calculation formula are converted into standard score. The total score of standard score ranges from 0 to 100, and the higher the score, the worse the quality of life [3].SF36 is a commonly used universal scale for the study of quality of life in patients with thyroid disease, which measures 8 health concepts and 1 self-rating of health changes.Eight of these health concepts are further divided into two categories, namely physical health and mental health.SF36 is a multi-item scale, each dimension contains 2 ~ 10 items, including a total of 36 items.The total score of SF36 is 100 points, and the higher the score, the better the health status [5].The purpose of this study was to evaluate the relationship between thyroid function and health-related quality of life (HRQOL) and related metabolic indicators in patients with hypothyroidism.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥18, ≤75 years old;
* clear diagnosis of primary hypothyroidism;
* Use the same dose of levothyroxine for ≥3 months;
* The levels of thyroid function (TSH, TT4, FT4, TT3, FT3) in hospital laboratory blood tests no more than 6 weeks before participation were within the normal range;

Exclusion Criteria:

* regnancy or lactation women
* affect blood sugar, blood lipid metabolism drugs
* serious heart disease
* thyroid malignant tumor
* history of mental illness

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hypothyroidism in Chaoyang Hospital outpatient department
Sampling Method: Non-Probability Sample
Enrollment: 98 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-11-01 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
Thyroid-specific Patient Reported Outcome(ThyPRO39) | 1year
  Correlation between thyroid function level and health-related quality of life (HRQOL) and metabolic indexes.

SECONDARY OUTCOMES:
the MOS 36-item Short Form Health Survey(SF36) | baseline
  Correlation between thyroid function level and health-related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Guang Wang, Principal Investigator — Beijing Chao-Yang Hospital, Capital Medical University, Beijing 100020, China
Locations (1):
- BeijingCYH, Beijing, Beijing Municipality, China